CLINICAL TRIAL: NCT01888887
Title: Cetaphil Daily Facial Cleanser: 200 Human Subject Repeat Insult Patch Test Skin Irritation/Sensitization Evaluation
Brief Title: Repeat Insult Patch Test of Skin Irritation/Sensitization for Cetaphil Daily Facial Cleanser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLI.04.SRE.US10236
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2013-06

CONDITIONS: Skin Irritation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetaphil Daily Facial Cleanser (Experimental): All subjects receive Cetaphil Daily Facial Cleanser
  Interventions: Other: Cetaphil Daily Facial Cleanser

INTERVENTIONS:
Other: Cetaphil Daily Facial Cleanser

SUMMARY:
Determine if Cetaphil Daily Facial Cleanser is a contact sensitizer or irritant to the skin

ELIGIBILITY:
Inclusion Criteria:

* Not currently under a doctor's care
* Free of dermatological or systemic disorder which would interfere with the results
* Free of any acute or chronic disease
* Will complete a preliminary medical history form and are in general good health
* Can read, understand, and sign informed consent

Exclusion Criteria:

* Under 18 years old
* Currently under doctor's care
* Currently taking any medication
* History of acute or chronic disease
* Diagnosed with chronic skin allergies
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
area of erythema and edema to test reaction of skin to product | 3 consecutive weeks
  9 consecutive 24hr exposures for every Monday, Wednesday, and Friday for 3 consecutive weeks will be conducted to test the reaction of the skin to the test product

CONTACTS AND LOCATIONS:
Overall Officials: Mayya Tastene, MD, Principal Investigator — AMA Laboratories
Locations (1):
- AMA Laboratories, New City, New York, United States